CLINICAL TRIAL: NCT07147751
Title: Characterization of Primary Central Nervous System Diffuse Large B Cell Lymphoma (PCNS-DLBCL) by Multiomic Approach
Status: Not yet recruiting | Type: Observational
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Other Study IDs: IELSG57
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Primary Central Nervous System Diffuse Large B Cell Lymphoma (PCNS-DLBCL)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Already existing and coded tumor biological material will be retrospectively collected from institutional biobanks upon receipt of ethical approval
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PCNS-DLBCL is a rare extranodal non-Hodgkin lymphoma that primarily affects the brain, spine, or vitreoretinal space. The prognosis for PCNS-DLBCL is significantly worse than that for its systemic counterpart.

Understanding how and where this tumor initiates, and how it survives or depends on the microenvironment of the CNS is key to understanding the underlying biology and identifying reliable biomarkers for selecting personalized therapy or for biologically directed therapy that could improve the cure rate of CNS lymphomas.

DETAILED DESCRIPTION:
Already existing and coded tumor biological material and health-related patient data will be retrospectively collected from institutional biobanks and patients' medical charts or electronic medical records upon receipt of ethical approval. Each patient enrolled in the study will be assigned a unique identification numerical code upon registration in the study. The unique identification code will be used to record health-related data and to label biological samples. The coded biological material will be transferred at the Institute of Oncology Research in Bellinzona and the IRCCS Policlinico San Matteo Foundation in Pavia.

Diagnostic slides will be centrally revised by a panel of expert pathologists to confirm the diagnosis of PCNS-DLBCL. Health-related data will be collected in the e-CRFs. Data quality will be ensured by query generation.

Annotated baseline features will include: age, sex, the date of diagnosis, ECOG PS, IELSG index, clinical features (i.e. neurologic signs or symptoms, psychiatric and behavioural changes, systemic lymphoma symptoms, and comorbidities), imaging features (i.e. MRI report), disease involvements (i.e. bone marrow infiltrate, CSF, Vitro-retinal, basal ganglia, corpus callosum, brain stem, or cerebellum), laboratory features (i.e. complete blood count parameters, LDH levels, HIV infection evidence, HCV infection evidence, HBV infection evidence, EBV infection evidence, CMV infection evidence, and cerebrospinal fluid examination parameters).

Annotated follow-up features will include: the start date, the regimen, the response level and the date of response evaluation of the first-line therapy, the start date, the regimen, the response level and the date of response evaluation of the second-line therapy; the date of transplantation and the date of relapse.

Survival features will include date of death, cause of death, and date of last follow-up.

All FFPE samples will undergo a comprehensive histological review, including immunohistochemical investigations aimed to analyze the various cell populations and the microenvironment; EBER ISH assay to verify the presence of latent EBV-infection, FISH assays to verify the presence of translocations involving BCL2, BCL6, and MYC genes, and of CDKN2A and 6p21-22 (HLA locus) loss.

Molecular analyses on tumor samples will include: 1) DNA alteration analysis by means of NGS approach; 2) genome-wide methylation profiling (the sole epigenetic fingerprints that can be robustly assayed on FFPE material); 3) transcriptional profiling; 4) Ig heavy chain (IGH) rearrangements detection and immunoglobulin heavy-chain variable region gene (IGHV) analysis.

The results of all these analyses will be recorded in the clinical-biological database. Statistical analysis will be performed to integrate and correlate obtained biological data with collected radiomic and clinical information, to outline a precise PCNS-DLBCL multiomic profile and to investigate unraveled genes or cellular pathways, potentially useful for diagnostic, predictive, and therapeutic purposes. Hierarchical clustering analysis will be performed to identify genetic driver alterations and discover any subsets of tumors with distinctive multiomic (genetic/transcriptomic/radiomic) signatures.

ELIGIBILITY:
Inclusion Criteria:

1. Be an adult immunocompetent patient who received a PCNS-DLBCL diagnosis according to the WHO-HAEM5 criteria between 2018 and 2024.
2. Availability of formalin-fixed paraffin-embedded (FFPE) diagnostic tumor material.
3. Availability of the baseline and follow-up annotations

Exclusion Criteria:

1. Established immunodeficiency conditions.
2. Secondary CNS localizations of DLBCL
3. Transformed DLBCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with primary central nervous system diffuse large B cell lymphoma (PCNS-DLBCL)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of non-GC phenotype | 12 months: from the end of samples collection to the end of study analysis
Prevalence of mutations, copy number abnormalities, and structural variants | 12 months: from the end of samples collection to the end of study analysis
Prevalence of PCNS-DLBCL molecular subtypes defined by genetic lesions | 12 months: from the end of samples collection to the end of study analysis
Prevalence of PCNS-DLBCL molecular subtypes defined by gene expression signatures | 12 months: from the end of samples collection to the end of study analysis
Prevalence of PCNS-DLBCL molecular subtypes defined by genetic methylation profile | 12 months: from the end of samples collection to the end of study analysis

SECONDARY OUTCOMES:
Prevalence of molecular features of clinical, laboratory, and radiological features | 12 months: from the end of samples collection to the end of study analysis
Prevalence of PCNS-DLBCL immunological signatures defined by gene expression profiling | 12 months: from the end of samples collection to the end of study analysis
3. Prevalence of PCNS-DLBCL MicroRNA signatures defined by miRNOMA evaluation | 12 months: from the end of samples collection to the end of study analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marco Paulli, MD, Study Chair — Unit of Pathology, IRCCS Policlinico San Matteo Foundation and Department of Molecular Medicine, University of Pavia (IT); Marco Lucioni, MD, Study Chair — Unit of Pathology, IRCCS Policlinico San Matteo Foundation and Department of Molecular Medicine, University of Pavia (IT)
Locations (2):
- Fondazione IRCCS Policlinico San Matteo Pavia, Pavia, Italy
- Oncology Institute of Southern Switzerland and Institute of Oncology Research, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No